# Hydroxychloroquine as Post-Exposure Prophylaxis Against COVID-19 Infection (PEPCOH)

# NCT04372017

Protocol Document including SAP

Continuing Review Date 03.11.2021

## **Protocol Title**

# <u>Post-Exposure Prophylaxis for COVID-19 with</u> <u>Hydroxychloroquine</u>

Protocol Number: **PEPCOH** 

Lead site Name: Sanford Health

Study Chair: Susan Hoover, MD

Version: 1.0 (2020.05.15)

NCT: 04372017

## Responsibility Acknowledgement:

I have read this study protocol and agree to adhere to the requirements. I will provide copies of this study protocol and all pertinent information to the study personnel. I will discuss this material with them and ensure they are fully informed regarding the study interventions and the conduct of the study according to the Food and Drug Administration (FDA) Guidelines for Good Clinical Practices (GCP), the institutional policies and procedures, and pertinent individual country laws/regulations.

| | Date |
|-----------------------------|------|
| Site Principal Investigator | |

## **Table of Contents**

| 1.0 | Protocol Summary | 6 |
|-----|------------------------------------------------------------------|----|
| 1.1 | Synopsis | 6 |
| 1.2 | Schema | 9 |
| 1.3 | Schedule of Activities (SoA) Cohort A & B | 10 |
| 2.0 | Introduction | 11 |
| 2.1 | Study Rationale | 11 |
| 2.2 | Background | 11 |
| 3.0 | Objectives and Endpoints | 11 |
| 3.1 | Primary Objectives | 11 |
| 3.2 | Primary Hypothesis: | 11 |
| 4.0 | Study Design | 12 |
| 4.1 | Overall study design | 12 |
| 4.2 | End of Study Definition | 12 |
| 5.0 | Study Population | 12 |
| 5.1 | Inclusion Criteria | 12 |
| 5.2 | Exclusion. | 12 |
| 5.2 | Screen Failures | 12 |
| 6.0 | Study Intervention | 12 |
| 6.1 | Study Intervention(s) Administered: | 12 |
| 6.2 | Hydroxychloroquine Sulfate (See Appendix C for more information) | 13 |
| 6.3 | Vitamin D with calcium (Cholecalciferol) | 16 |
| 6.4 | Participant Implications | 17 |
| 6.5 | Drug Inventory Records | 18 |
| 6.6 | Measures to Minimize Bias: Randomization and Blinding | 18 |
| 6.7 | Study Intervention Compliance | 18 |
| 6.8 | Concomitant Therapy | 18 |
| 6.9 | Intervention after the End of the Study | 18 |
| 7.0 | Participant Discontinuation/Withdrawal | 18 |

| 7. | 1 1 | Discontinuation of Study Intervention: | 19 |
|------|-------|--------------------------------------------|----|
| 7.2 | 2 I | Participant Withdrawal from the Study | 19 |
| 7.3 | 3 I | Lost To Follow Up | 19 |
| 8.0 | Stu | dy Procedures and Safety Assessments | 20 |
| 8. | 1 A | Administrative Procedures | 20 |
| | 8.1.1 | Screening Procedures | 20 |
| | 8.1.2 | Informed Consent | 20 |
| | 8.1.3 | Inclusion/Exclusion Criteria | 21 |
| | 8.1.4 | Assignment of Screening Number | 21 |
| | 8.1.5 | Enrollment | 21 |
| | 8.1.6 | Assignment of Study Participant Number | 21 |
| 8.2 | 2 ( | Clinical Procedures/Assessments | 21 |
| | 8.2.1 | Participant Reported Outcomes | 21 |
| | 8.2.2 | Adverse Event (AE) Monitoring | 22 |
| 8.3 | 3 A | Adverse events and Serious Adverse Events: | 22 |
| | 8.3.1 | AE and SAE Collection and Reporting | 23 |
| | 8.3.2 | AE/SAE Assessments | 23 |
| | 8.3.3 | Safety Review Committee (SRC) | 24 |
| 9.0 | Sta | tistical Considerations | 24 |
| 9. | 1 5 | Statistical Hypothesis | 24 |
| 9.2 | 2 5 | Sample Size Determination | 24 |
| 9.3 | 3 5 | Statistical Analyses | 25 |
| 9.4 | 4 I | nterim Analysis | 25 |
| 10.0 | Reg | gulatory, Ethical, and Study Oversight | 26 |
| 10 | .1 \$ | Statement of Compliance | 26 |
| 10 | .2 I | nformed Consent | 26 |
| 10 | .3 | Study Participant Confidentiality | 27 |
| 10 | .4 I | Risks and Benefits | 27 |
| 10 | .5 I | Ethics | 27 |

| | 10.6 | Study Documentation and Case Report Forms (CRFs) | 27 |
|----|---------|--------------------------------------------------|----|
| | 10.7 | Document and Data Retention | 28 |
| | 10.8 | Direct Access to Source Data/Documents | 28 |
| | 10.9 | Protocol Compliance | 28 |
| | 10.10 | Publication Policy | 28 |
| Aj | ppendix | A: Abbreviations | 29 |
| Aj | ppendix | B: Protocol Amendment History | 30 |
| Aj | ppendix | C: Hydroxychloroquine Drug Information | 31 |
| Aj | ppendix | CD: Exclusion Medication List | 33 |
| Αį | ppendix | x E: References | 50 |

## 1.0 Protocol Summary

## 1.1 Synopsis

| Title of Study | Post-Exposure Prophylaxis for COVID-19 with Hydroxychloroquine (PEPCOH) |
|---|---|
| Study Objectives | <ul> <li><u>Cohort A:</u> Determine whether post-exposure prophylaxis with hydroxychloroquine can prevent COVID-19 in healthcare workers who have been exposed to a known case of COVID-19.</li> <li><u>Cohort B:</u> Determine whether post-exposure prophylaxis with hydroxychloroquine can prevent COVID-19 in high-risk individuals who have been exposed to a known case of COVID-19.</li> <li>Primary Hypothesis:</li> </ul> |
| | <ul> <li><u>Cohort A:</u> Primary Hypothesis: Hydroxychloroquine will reduce the number of healthcare workers that convert to infected status post-exposure compared with placebo.</li> <li><u>Cohort B:</u> Primary Hypothesis: Hydroxychloroquine will reduce the number of high-risk individuals that convert to infected status post-exposure compared with placebo.</li> </ul> |
| Study Design | A multi-cohort, prospective, double-blind, randomized, placebo controlled study |
| <b>Study Population</b> | <ul> <li>Inclusion Criteria Cohort A:</li> <li>≥ 18 years old</li> <li>Employee of healthcare organization in South Dakota or Sanford Health employee in any location and with exposure to a person with COVID-19 within the last 5 days</li> <li>Occupational exposure as determined by the participant's employee health department (i.e. not wearing the proper Personal Protective Equipment (PPE))</li> <li>Criteria according to Center for Disease Control (CDC) guidelines</li> <li>Community exposure (within 6 feet for at least 15 minutes)</li> <li>No current symptoms attributable to COVID-19, per HCW report (fever, cough, difficulty breathing, sore throat)</li> <li>No prior COVID-19 positive diagnosis (eligible if previous testing is negative and meets all other inclusion and exclusion)</li> <li>Ability to provide informed consent</li> </ul> |
| | <ul> <li>Inclusion Criteria – Cohort B</li> <li>≥ 18 years old</li> <li>High-risk person who had close contact (i.e. within 6 feet for at least 15 minutes) with a COVID-19 positive person within the last 5 days and is a South Dakota resident or high-risk person with close household contact of a COVID-19 positive Sanford employee</li> </ul> |

- High-risk person defined by:
  - Age 18-44 with 2 or more comorbidities listed below
  - Age 45-79 with any comorbid condition listed below
  - Age 80 and above (regardless of comorbid conditions)
  - Co-morbid list
    - o Congestive Heart Failure (CHF)
    - Chronic lung disease<sup>¥</sup>
    - Solid organ transplant or immunosuppression\*
    - o Chronic Kidney Disease or End Stage Renal Disease
    - Diabetes mellitus
    - o Cardiovascular disease/Hypertension
    - o Smoking/Vaping (currently using or history of using in the past 1 year)
    - Obesity (calculated by height and weight per participant report)
    - Hyperlipidemia
    - ¥ Includes any of the following: asthma, chronic obstructive pulmonary disease, emphysema
    - \* Defined as an outpatient prescription of greater than 10 mg/day of prednisone or equivalent, use of chemotherapy, or use of immunosuppressive agents for solid organ transplant or for an autoimmune disease.
- No current symptoms attributable to COVID-19
- No prior COVID-19 positive diagnosis (eligible if previous testing is negative and meets all other inclusion and exclusion)
- Ability to provide informed consent
- Confirmed review of concomitant medications (with emphasis on cardiac medications)

#### **Exclusion Criteria:**

#### **Exclusion Criteria Cohort A & B:**

- Known allergy to hydroxychloroquine or quinine
- Known history of long QT syndrome
- Known history of arrhythmia or dysrhythmia
- Known current QTc >500 ms
- Known G6PD deficiency
- Known history of hypoglycemia
- Pregnant or Nursing by patient history
- Use of any of the following concomitant medications: See Appendix D for Exclusion medication list
- Concurrent diagnosis of dermatitis, porphyria, or psoriasis
- History of chronic liver disease, including cirrhosis and/or diagnosis of hepatitis (infectious, idiopathic, or immune)
- History of chronic kidney disease
- Pre-existing retinopathy
- Already taking hydroxychloroquine
- Any condition or medication in the opinion of the investigator that would prohibit the use of hydroxychloroquine
- Enrollment in another clinical with investigational drug or device
- Inability to swallow pills
- Adults unable to provide informed consent

| Sample Size | Cohort A n= 1356 |
|---|---|
| | Cohort B n= 383 |
| Study<br>Intervention | Hydroxychloroquine vs. Placebo (Vitamin D with calcium) |
| Study<br>Evaluations | Assessments on this study will be completed as outlined in Section 8.3. |
| Study Period | Planned start date: April 2020 Planned accrual start date: April 2020 Planned accrual closure: April 2021 Planned study closure: April 2022 |

## 1.2 Schema



9

## 1.3 Schedule of Activities (SoA) Cohort A & B

This study consists of screening, enrollment and randomization, treatment, and follow-up. Follow-up will include evaluation of the treatment and subsequent infection, re-infection, adverse events, and long-term sequelae of treatment and/or infection. The detailed schedule of study procedures and assessments with the time intervals is shown in Table 1.

Table 1

| | Screening | & Enrollment | Treatment / Placebo Phase | | | Follow-up <sup>b</sup> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening <sup>a</sup> | Enrollment /<br>Randomization | Day 1 | Day 2 | Day 3f | Day 4 | Day 5 | Day 14<br>( <u>+</u> 1 day) | Day 35 <sup>e</sup><br>(+3 days) | 12 Months<br>( <u>+</u> 30 days) |
| Informed Consent /<br>HIPAA | X | | | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | | | |
| Demographics | X | | | | | | | | | |
| Randomization | | X | | | | | | | | |
| Hydroxychloroquine /<br>Placebo (Vitamin D with<br>calcium) | | | X | X | X | X | X | | | |
| Patient Reported symptoms <sup>c</sup> | | | | | X | | X | X | X | |
| Adverse Event<br>Assessment | | | | | X | | X | X | X | X |
| Outcomes <sup>d</sup> | | | | | | | | X | X | X |

a. Screening must be completed within 48 hours prior to study enrollment

b. Follow-up visits will consist of a phone call to the patient. Hydroxychloroquine and placebo patients will be followed.

c. Includes: patient reported temperature, cough, difficulty breathing, sore throat, chills, muscle pain, headache, new loss of taste or smell, and diarrhea.

d. Did the patient acquire COVID-19?

e. Day 35 should be at least 30 days (+3 days) post last dose of drug.

f. Day 3 and 5 AE assessment via phone call. (window ±1day)

#### 2.0 Introduction

#### 2.1 Study Rationale

Currently, prevention of person-to-person transmission of SARS-CoV-2, the virus which causes COVID-19, is achieved by reducing close contact through physical distancing measures and through the use of personal protective equipment (PPE) in the healthcare setting. The effect of post-exposure medication treatment on acquisition of infection or progression to symptomatic disease is unknown.

#### 2.2 Background

Coronavirus Infectious Disease-2019 (COVID-19) is an infection caused by a novel virus, Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), which emerged in the winter of 2019 initially in China, then spread to involve the entire world in a pandemic. Infected individuals may be asymptomatic, while others demonstrate a range of symptoms from upper respiratory symptoms to pneumonia, respiratory failure, acute respiratory distress syndrome, or death. Hydroxychloroquine inhibits SARS-CoV-2 replication in vitro and may have antiviral effects in people with COVID-19 disease (Yao *et al.* 2020). It is postulated that early preemptive therapy may prevent disease or reduce severity, but its effectiveness in the

## 3.0 Objectives and Endpoints

## 3.1 Primary Objectives

post-exposure setting is unknown.

- <u>Cohort A:</u> Determine whether post-exposure prophylaxis with hydroxychloroquine can prevent COVID-19 in healthcare workers with direct patient contact who have been exposed to a known case of COVID-19.
- <u>Cohort B:</u> Determine whether post-exposure prophylaxis with hydroxychloroquine can prevent COVID-19 in high-risk individuals who have been exposed to a known case of COVID-19.

#### 3.2 Primary Hypothesis:

- <u>Cohort A:</u> Primary Hypothesis: Hydroxychloroquine will reduce the number of healthcare workers that convert to infected status post-exposure compared with placebo.
- <u>Cohort B:</u> Primary Hypothesis: Hydroxychloroquine will reduce the number of high-risk individuals that convert to infected status post-exposure compared with placebo.

## 4.0 Study Design

#### 4.1 Overall study design

This is a prospective, double-blind, randomized, placebo-controlled study in two distinct cohorts to evaluate the efficacy and safety of hydroxychloroquine in the prevention of COVID-19 infection. Additional sub-studies will be added and removed throughout this larger "tent" protocol to answer other objectives. These studies will be listed in the appendices of this protocol.

Other non-Sanford institutions will be allowed to participate in this study after all legal and regulatory documents are final.

Sanford Health will function as the lead site for trial oversight.

#### 4.2 End of Study Definition

A participant is considered to have completed the study if he/she has completed all phases of the study including last follow up visit at 12 months.

## 5.0 Study Population

#### 5.1 Inclusion Criteria

See Synopsis (section 1.1)

#### 5.2 Exclusion

See Synopsis (section 1.1)

#### 5.2 Screen Failures

Screen failures are defined as participants who consent to participate in the clinical study but are not subsequently enrolled. A minimal set of screen failure information is required to ensure transparent reporting of screen failure participants. Minimal information should include demography, screen failure details, eligibility criteria, and any serious adverse event (SAE). Screen failures will not count towards total enrollment.

## 6.0 Study Intervention

#### **6.1** Study Intervention(s) Administered:

Hydroxychloroquine/placebo (vitamin D with calcium) will be administered as part of this study. Randomization will occur at a 1:1 ratio in each cohort. Participation in additional non-interventional clinical research studies is allowed. If the participant becomes infected with COVID-19, the participant will stop the intervention and be treated per the discretion of their primary care provider.

Subjects enrolled will be assigned to the appropriate cohort and randomized to receive hydroxychloroquine 200mg tablets, Day 1-2 tablets by mouth twice per day, Day 2-5 1 tablet by mouth twice per day (total of 12 tablets) or placebo. Placebo will be vitamin D with calcium tablets 10mcg tablet - Day 1-2 tablets by mouth twice per day, Day 2-5 1 tablet by mouth twice per day (total of 12 tablets). Subjects will be monitored for any toxicities during and after treatment.

**Table 2. Intervention dosing** 

| Drug | Dose | Dose Frequency | Route |
|---|---|---|---|
| Hydroxychloroquine | 2 tablets | Twice daily on day 1 | PO |
| 200 mg tablets | 1 tablet | Twice daily on days 2-5 | PO |
| Placebo (vitamin D with calcium, | 2 tablets | Twice daily on day 1 | PO |
| 10mcg/25mg tablets) | 1 tablet | Twice daily on days 2-5 | PO |

## 6.2 Hydroxychloroquine Sulfate (See Appendix C for more information)

#### 6.2.1. Other Names

IUPAC: 2-[4-[(7-chloroquinolin-4-yl)amino]pentylethylamino]ethanol

MeSH: Plaquenil; Hydroxychlorochin; Hydroxychloroquine; Hydroxychloroquine Sulfate: Hydroxychloroquine Sulfate (1:1) Salt; Oxychlorochin; Oxychloroquin; 4-aminoquinoline

#### 6.2.2. Classification

Immunosuppressive, anti-inflammatory, anti-autophagy, and anti-malarial

#### 6.2.3. Dose Specifics

One tablet of 200 mg of hydroxychloroquine sulfate is equivalent to 155 mg base. See section 6.1 for dosing.

#### 6.2.5. Preparation

No special preparation.

#### 6.2.6. Administration

Take hydroxychloroquine sulfate by mouth, preferably with a meal or a glass of milk.

#### 6.2.7. Contraindications

Use of hydroxychloroquine sulfate is contraindicated in patients with known hypersensitivity to 4-aminoquinoline compounds. Use with

caution in patients with alcoholism, hepatic/renal dysfunction, glucose-6-phosphate dehydrogenase (G-6-PD) deficiency, gastrointestinal, neurological, or blood disorders. A dose reduction may be required.

#### 6.2.8. Availability

Commercially available as a tablet for oral administration. For the purposes of this study the tablet drug will be provided by Sanford Research and supplied in 200mg tablets with matching placebo.

#### 6.2.9. Side Effects

#### 1. Ocular:

It is recommended that hydroxychloroquine be discontinued if ocular toxicity is suspected and the patient should be closely observed given that retinal changes (and visual disturbances) may progress even after cessation of therapy.

Retinal toxicity from hydroxychloroquine is serious but very rare. The incidence rises sharply to about 1% at 5 years of use, so the American Academy of Ophthalmology recommends screening starting after 5 years. Toxicity is more common with doses exceeding 400 mg/day or a total dose of more than 1000 g. This study dose is 800 mg for 1 day then 400 mg for 4 more days (Marmor *et al.* 2011).

2. <u>Cardiac</u>: Post marketing cases of life-threatening and fatal cardiomyopathy have been reported with use of hydroxychloroquine sulfate. Patients may present with atrioventricular block, pulmonary hypertension, and sick sinus syndrome or with cardiac complications. Electrocardiogram (ECG) findings may include atrioventricular, right or left bundle branch block. Signs or symptoms of cardiac compromise have appeared during acute and chronic treatment. Clinical monitoring for signs and symptoms of cardiomyopathy is advised. Chronic toxicity should be considered when conduction disorders (bundle branch block/atrio-ventricular heart block) or biventricular hypertrophy are diagnosed. If cardiotoxicity is suspected, prompt discontinuation of hydroxychloroquine sulfate may prevent life-threatening complications.

Hydroxychloroquine sulfate prolongs the QT interval. Ventricular arrhythmias and torsades de pointes have been reported in patients taking hydroxychloroquine. Therefore, hydroxychloroquine sulfate should not be administered with other drugs that have the potential to prolong the QT interval.

Hydroxychloroquine has been used for decades for malaria and autoimmune disease without pre-treatment EKGs or routine cardiac monitoring. A 2018 review of short-term antimalarial treatment including chloroquine, which is known to carry greater risk of toxicity, found no serious cardiac adverse events among participants (n=1076), receiving acute therapy for malaria. With chronic use of hydroxychloroquine (years), QT prolongation and cardiomyopathy have occurred. This study uses a 5-day course and subjects with heart disease will be excluded (Haeusler et al. 2018).

- 3. Worsening of Psoriasis and Porphyria: Use of hydroxychloroquine sulfate in patients with psoriasis may precipitate a severe attack of psoriasis. When used in patients with porphyria the condition may be exacerbated. The preparation should not be used in these conditions unless in the judgment of the physician the benefit to the patient outweighs the possible hazard.
- 4. Proximal Myopathy and Neuropathy: Skeletal muscle myopathy or neuropathy leading to progressive weakness and atrophy of proximal muscle groups, depressed tendon reflexes, and abnormal nerve conduction, have been reported. Muscle and nerve biopsies have been associated with curvilinear bodies and muscle fiber atrophy with vacuolar changes. Assess muscle strength and deep tendon reflexes periodically in patients on long-term therapy with hydroxychloroquine sulfate.
- 5. <u>Neuropsychiatric Events, Including Suicidality:</u> Suicidal behavior has been rarely reported in patients treated with hydroxychloroquine sulfate.
- 6. <u>Hypoglycemia</u>: Hydroxychloroquine sulfate has been shown to cause severe hypoglycemia including loss of consciousness that could be life threatening in patients treated with or without antidiabetic medications. Patients treated with hydroxychloroquine sulfate should be warned about the risk of hypoglycemia and the associated clinical signs and symptoms. Patients presenting with clinical symptoms suggestive of hypoglycemia during treatment with hydroxychloroquine sulfate should have their blood glucose checked and treatment reviewed as necessary.
- 7. <u>Dermatologic Effects:</u> Dermatologic reactions to hydroxychloroquine sulfate may occur and, therefore, proper care should be exercised when it is administered to any patient receiving a drug with a significant tendency to produce dermatitis.

#### 6.3 Vitamin D with calcium (Cholecalciferol)

6.3.1 Other Names IUPAC Name: (1S,3Z)-3-[(2E)-2-[(1R,3aS,7aR)-7a-methyl-1-[(2R)-6-methylheptan-2-yl]-2,3,3a,5,6,7-hexahydro-1H-inden-4-ylidene]ethylidene]-4-methylidenecyclohexan-1-ol

MeSH: (3 beta,5Z,7E)-9,10-Secocholesta-5,7,10(19)-trien-3-ol; Calciol; Cholecalciferol; Vitamin D3

- 6.3.2 Classification Lipophilic secosteroid
- 6.3.3 Mode of Action

Vitamin D with calcium is dietary supplement used to promote calcium absorption in intestines, bone resorption, increase phosphate levels to maintain skeletal calcium balance. *In vivo* synthesis of the major biologically active metabolites of vitamin D with calcium occurs in two steps. First, in the liver microsomal enzymes convert vitamin D to calcifediol (25-hydroxycholecalciferol). Second, calcifediol is released into systemic circulation where it binds vitamin D-binding protein, an α-globulin carrier protein that transports it to the proximal tubules of the kidneys where Parathyroid hormone regulates its further hydroxylation to calcitriol (1,25-dihydroxycholecalciferol). Calcitriol is again released into systemic circulation, binds to vitamin D-binding protein and is distributed to throughout the body including to target organs like intestine, kidney, and bone. Vitamin D is indicated in treatment of hypoparathyroidism, refractory rickets, and familial hypophosphatemia.

Vitamin D3 and vitamin D2 are bioequivalent.

#### 6.3.4 Storage and Stability

Vitamin D3 with calcium tablets are stored at room temperature 15°-30°C (59°-86°F), protect from light and moisture. They should be dispense in a tight, light-resistant container.

6.3.5 Dose Specifics

Placebo will be vitamin D with calcium tablets 10mcg/25mg tablet. See section 6.1 for dosing.

6.3.6 Preparation

No special preparation.

6.3.7 Administration

Take Vitamin D3 with calcium by mouth with meal or a glass of milk.

Take hydroxychloroquine sulfate by mouth, preferably with a meal or a glass of milk.

#### 6.3.8 Contraindications:

Use of Vitamin D3 with calcium is contraindicated in patients with renal impairment, heart disease, kidney stones, arteriosclerosis, and individuals with hypercalcemia, hypervitaminosis D; gastrointestinal, liver, or biliary disease associated with malabsorption of vitamin D analogues and drugs that could have allergenic cross reactivity/hypersensitivity with Vitamin D3.

#### 6.3.9 Availability

Commercially available as a tablet for oral administration. For the purposes of this study the tablet drug will be provided by Sanford Research and supplied in 10mcg/25mg tablets as placebo.

#### 6.3.10 Side Effects

- 1. <u>Renal:</u> Impairment of renal function with polyuria, nocturia, polydipsia, hypercalcemia, reversible azotemia, hypertension, nephrocalcinosis, generalized vascular calcification, or irreversible renal insufficiency which may result in death
- 2. <u>Central Nervous System (CNS)</u>: Mental retardation, disorientation, confusion
- 3. <u>Soft Tissues</u>: widespread calcification of the soft tissues, including the heart, blood vessels, renal tubules, and lungs
- 4. <u>Skeletal:</u> Bone demineralization (osteoporosis) in adults. Decline in the average rate of linear growth and increased mineralization of bones in infants and children (dwarfism), vague aches, stiffness, and weakness
- 5. Gastrointestinal: Nausea, anorexia, and constipation
- 6. Metabolic: Mild acidosis, anemia, and weight loss
- 7. <u>Teratogenic effects:</u> supravalvular aortic stenosis, elfin facies, and mental retardation recorded in pregnant women with hypervitaminosis D

### 6.4 Participant Implications

- 1. If a participant vomits after taking their dose study drug it will be considered a missed dose and not retaken. The participant will resume with the next scheduled dose.
- 2. If the participant forgets to take a dose, that dose will not be made up and participant will resume with the next scheduled dose.
- 3. If the participant is unable to start the hydroxycholoroquine / vitamin D with calcium in the morning on Day 1 due to delivery timing, the participant is allowed to initiate Day 1 with an evening dose.
- 4. Participants should have at least 8 hours between doses.

5. Participants will be instructed to inform the study coordinator of any medication changes while on the active phase of the study

#### 6.5 Drug Inventory Records

Investigational Product Records at Investigational Site(s): It is the responsibility of the Investigator to ensure that a current record of investigational product disposition is maintained at each study site where investigational product is inventoried and disposed.

#### 6.6 Measures to Minimize Bias: Randomization and Blinding

On enrollment day, the participant will be assigned a unique number (randomization number). The randomization number encodes the participant's assignment to hydroxychloroquine or placebo (vitamin D with calcium), according to the randomization schedule generated prior to the study by the Sanford Command Core. Each participant will be dispensed randomized study intervention, labeled with his/her unique randomization number, throughout the study.

In the event of a Quality Assurance audit, the auditor(s) will be allowed access to study intervention records at the site(s) to verify that randomization/dispensing has been done accurately.

#### **6.7** Study Intervention Compliance

A pill diary will be given to each enrolled participant to document pill compliance.

## 6.8 Concomitant Therapy

- See inclusion and exclusion criteria for medications that are not allowed.
- No washout period is needed for hydroxychloroguine.
- Vaccines are allowed while on the study.

## 6.9 Intervention after the End of the Study

Participants who acquire COVID-19 while on study intervention as determined by a positive test indicating COVID-19 will be instructed to discontinue the study intervention by the study team. Participants will be unblinded and subsequent treatment will be at the discretion of their primary care physician or provider who ordered the COVID-19 testing.

## 7.0 Participant Discontinuation/Withdrawal

Participants may withdraw consent at any time for any reason or be withdrawn from the trial at the discretion of the investigator should any untoward effect occur. In addition, a participant may be withdrawn by the investigator if enrollment into the trial is inappropriate, the trial plan is violated, or for administrative and/or other safety reasons.

#### 7.1 Discontinuation of Study Intervention:

A participant must be discontinued from the trial for any of the following reasons:

- The participant withdraws consent.
- Intercurrent illness that prevents further administration of treatment
- The participant has a confirmed positive pregnancy test
- The participant is lost to follow-up

At the discretion of the investigator for safety, behavioral, compliance, or administrative reasons.

For those participants who discontinue study intervention early, each participant will be followed for 30 days for acute adverse event monitoring.

## 7.2 Participant Withdrawal from the Study

- A participant may withdraw from the study at any time at his/her own request, or may be withdrawn at any time at the discretion of the investigator for safety, behavioral, compliance, or administrative reasons.
- If the participant withdraws consent for disclosure of future information, any data collected be for that time may be retained.

### 7.3 Lost To Follow Up

All reasonable efforts must be made to locate participants to determine and report their ongoing status. This includes follow-up with persons authorized by the participant.

Lost to follow-up is defined by:

- The inability to reach the participant after a minimum of two documented phone calls and
- Lack of response by participant to one certified mail letter.

All attempts should be documented in the participant medical record. Should the participant continue to be unreachable, he/she will be considered lost to follow up. Outcome information that is available via electronic medical records will be documented if available.

If it is determined that the participant has died, the site will use permissible local methods to obtain the date and cause of death.

## 8.0 Study Procedures and Safety Assessments

#### **8.1** Administrative Procedures

#### **8.1.1** Screening Procedures

All participants must agree to participate in the study prior to any study specific screening procedures being performed. Every participant shall be provided an Institutional Review Board (IRB)-approved informed consent to review and keep for his/her records.

Once consent has been documented, the site will assign the participant a screening number. A Screening Log of consented patients will be maintained at each site.

Screening evaluations will be used to determine the eligibility of the participant for study inclusion. All screening activities must be completed within 48 hours prior to study enrollment and include the following:

- Inclusion/Exclusion Criteria
- Demographics and Medical History

All screening evaluations must be completed and reviewed by the site investigator or healthcare licensed designee to confirm that potential participants meet all eligibility criteria. The study team will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

#### 8.1.2 Informed Consent

A study team member must obtain documented consent from each potential participant prior to participating in a clinical trial. This study will utilize an electronic consent process based in REDCap, a CFR part 11 compliant research database. An electronic version of the informed consent form will be approved by the IRB prior to use. When a participant is contacted for enrollment into the study, an email containing a unique link will be generated by REDCap and sent to the patient while on the phone with a study team member. A password will be provided to the participant verbally over the phone that is required to access the informed consent. This provides confirmation of the identity of the participant. Once the informed consent form has successfully accessed, the study team member will allow a period of time of 1-4 hours for the participant to read the informed consent and formulate questions. The study team member will place another call with the participant and proceed to have an informed consent discussion, answering any questions the participant might have. If the participant is willing to participate in the study, he or she will proceed to provide an electronic signature using a mouse or their finger and save the document. This locks the document from any further changes. An email containing a copy of the signed informed consent form will be generated via REDCap and emailed to the participant. A PDF of the signed informed consent document will be saved in the participant's medical record as well as printed out for the study file.

A copy of the consent form will be automatically generated via REDCap and emailed to the participant before participation in the trial. The research team member who obtained consent will record the consenting process per their institutional guidelines.

The initial informed consent form, any subsequent revised written informed consent form and any written information provided to the participant must receive the IRB's approval in advance of use. The participant will be informed in a timely manner if new information becomes available that may be relevant to the participant's willingness to continue participation in the trial. The informed consent will adhere to IRB requirements, applicable laws and regulations.

#### 8.1.3 Inclusion/Exclusion Criteria

All inclusion and exclusion criteria will be reviewed by the site Principal Investigator (PI) or licensed designee to ensure that the participant qualifies for the study.

#### 8.1.4 Assignment of Screening Number

Consented participants will be assigned a screening number.

#### 8.1.5 Enrollment

Once all screening procedures have been completed the site PI or licensed designee (RN, CNP, pharmacist, or physician) on the study team will review acknowledge the inclusion/exclusion source document. If the potential participant is determined to be eligible, the study site will enroll the participant in appropriate cohort in the electronic data capture (EDC) and then randomized by the Sanford Command Core to the intervention assignment. Sites will be notified by email in real time the randomization confirmation. The site study team will maintain an enrollment log and the lead site will maintain a study-wide enrollment log. If the potential participant is not eligible and becomes a screen fail, the reason will be noted on the inclusion/exclusion in the EDC and filed in the study records.

#### 8.1.6 Assignment of Study Participant Number

Participants will be assigned a participant study number at enrollment at the same time as randomization by the EDC. This number will be unique to this participant.

#### 8.2 Clinical Procedures/Assessments

See Schedule of events for activities that need to be done at each visit.

#### 8.2.1 Participant Reported Outcomes

Participant self-reported COVID-19 symptoms (temperature, cough, difficulty breathing, and sore throat) will be collected by the study team at time points outlined in the SoA. Participants will also be asked if they have or are

currently experiencing any other symptoms since starting the study intervention. These will be included in the adverse event monitoring.

#### 8.2.2 Adverse Event (AE) Monitoring

The investigator or licensed designee (RN, CNP, pharmacist, or physician) on the study team will assess each participant to evaluate for potential new or worsening AEs as specified in the SoA and more frequently if clinically indicated. If participant reported symptoms are an AE, the event will be tracked as an AE.

Participants will be followed and accessed for acute AEs until day 35 (30 days after the last dose of study medication). AEs will be documented accordingly. Adverse events will also be assessed at the 12 month follow up visit.

#### 8.3 Adverse events and Serious Adverse Events (SAE):

An AE is defined as any untoward or unfavorable medical occurrence in human participants, including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether considered related to the participant's participation in the research or not. AEs encompass both physical, psychological harms, and biochemical abnormalities. AEs may be reported by the participant, observed by the Investigator, or documented in medical records.

The site investigator and any licensed designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study intervention or study procedures, or that caused the participant to discontinue the study treatment. The site investigator or licensed designee will evaluate all adverse events according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. Toxicities will be characterized in terms regarding grade (seriousness), causality/attribution (see section 8.3.2), and action taken with regard to trial intervention.

Any adverse event which changes CTCAE grade over the course of a given episode will have each change of grade recorded on the adverse event case report forms/worksheets.

If the adverse event meets any of the criteria below, it is regarded as a SAE:

- the event led to the death of the participant
- the event led to serious deterioration in the health of the participant, that either resulted in:
  - o a life-threatening illness or injury
  - o a permanent impairment of a body structure or a body function
  - o in-patient or prolonged hospitalization

• an important medical event- defined as an event requiring medical or surgical intervention to prevent one of the outcomes listed above in this definition.

### 8.3.1 AE and SAE Collection and Reporting

All acute SAEs/AEs will be collected from the time the informed consent form (ICF) is signed until day 35. Follow-up of AEs will end either when the symptom or illness resolves completely, up to 30 days past the end of study participation (if ongoing at the time of study exit) or until the investigator determines that the event has stabilized and will not completely resolve. Participants will be assessed at the 12 month visit for any potential adverse events that could be attributable to hydroxychloroquine.

AEs to be reported include:

- All SAEs regardless of attribution
- All Cardiac AEs for Grade 2 and above that are attributed to intervention (possible, probable, and definite)
- All AEs grade 3 and above regardless of attribution

# Enrollment will be held and the SRC committee will meet if the following occur:

- Any SAEs with an attribution of possible, probable, and definite
- Any Cardiac AEs for Grade 2 and above that are attributed to intervention (possible, probable, and definite)
- Any AEs grade 3 and above attributed to intervention (possible, probable, and definite)

The SRC will review safety data and determine if the study can continue.

#### 8.3.2 AE/SAE Assessments

All AE and SAE reporting will be conducted in compliance Sanford Health Policy HRP 024 New Information.

AE assessments will be focused on body systems with potential known toxicities and well as other toxicities verbalized by the participant.

All AE and SAEs will be assigned causality by the Investigator in their relationship to the study medication based on the following categories:

- <u>Definitely:</u> clear evidence exists that the event was caused by the intervention
- <u>Probably:</u> reasonable probability exists that the event was caused by the intervention
- <u>Possibly:</u> reasonable possibility exists that the event may have been caused by the intervention
- <u>Unlikely:</u> evidence exists that the event was caused by other factors; although the relationship of the event to the intervention cannot be completely ruled out, is remote

• <u>Unrelated:</u> the cause of the event is known and the event is in no way related to any aspect of the intervention

SAEs must be reported to the lead site and study chair at <a href="SH\_HCQ\_Team@sanfordhealth.org">SH\_HCQ\_Team@sanfordhealth.org</a> as soon as possible, but no later than 24 hours from the day the study team became aware of the event. Follow-up reports may be required or requested by the lead site or regulatory agency and should be completed promptly.

IRB notification of SAEs is required per Sanford IRB reporting guidelines. Investigators and study personnel are responsible for knowing IRB reporting requirements. Reporting of SAEs, whether related or unrelated to the study participation, should follow the most stringent rules for reporting.

The date of onset of the event, the date the site staff became aware of the event and determined it met the criteria of an SAE, and the date the event resolved or no longer fit the criteria of SAE will be documented in the source document and in the EDC system.

#### 8.3.3 Safety Review Committee (SRC)

An independent SRC will be established with experienced members, none of whom are participating as study investigators, to monitor and evaluate the safety of subjects, to maintain oversight of study data and to monitor progress of the study. The committee will initially meet monthly and more frequently if concerns of safety are noted. The findings of the SRC will be submitted to the IRB within 10 days after the meeting. All SAEs will be reported to the SRC as soon as possible after learning of the event.

The Study Chair will review cumulative AEs and SAEs weekly and will share concerns with the SRC. The SRC will make recommendations to the Study Chair regarding steps to ensure subject safety and the continued ethical integrity of the trial. The SRC will review interim study results and consider the overall risk and benefit to trial participants. The SRC will recommend to the Study Chair whether the trial should continue in accordance with the protocol.

### 9.0 Statistical Considerations

#### 9.1 Statistical Hypothesis

There will be a 50% decrease (relative risk reduction) in the conversion to infected status within the treatment arm compared to the control arm.

### 9.2 Sample Size Determination

#### Cohort A:

It is expected that 10% of exposed healthcare workers will convert to infected status without intervention. The treatment arm will be assumed to have a conversion of 5% (50% relative reduction, 5% absolute risk reduction). Due to the uncertainty of this

trial, a conservative 10% drop out rate is included in the calculation. Under these assumptions (Treatment: 5% infected, Control: 10% infected,  $\alpha$ : 0.0492, Power: 90%), the total sample size is 1356 patients (610 patients are needed in each arm + 10% dropout = 1356 total patients).

#### Cohort B:

It is expected that 30% of exposed high risk patients will convert to infected status without intervention. The treatment arm will be assumed to have a conversion of 15% (50% relative reduction, 15% absolute risk reduction). Due to the uncertainty of this trial, a conservative 10% drop out rate is included in the calculation. Under these assumptions (Treatment: 15% infected, Control: 30% infected,  $\alpha$ : 0.0492, Power: 90%), the total sample size is 383 patients (172 patients are needed in each arm + 10% dropout = 383 total patients).

#### 9.3 Statistical Analyses

All baseline and demographic variables such as race, gender, age, height, and weight will be summarized. Continuous variables will be summarized using mean, standard deviation, median, IQR, minimum and maximum. Categorical variables will be presented using frequencies and percentages.

Difference in infected status proportions between the treatment and control groups will be evaluated using Fisher's exact test. The number of adverse events, rate of occurrence, and severity by treatment group will be reported and statistically compared using non-parametric methods.

Details of the analysis methods will be provided in the Statistical Analysis Plan (SAP), which will be finalized as early as possible after enrollment commences in order to minimize bias in the analysis strategy.

#### 9.4 Interim Analysis

An interim analysis will be conducted to determine if the study should be stopped due to safety concerns or efficacy. Using O'Brien-Fleming approach, the interim analysis will use a significance level of  $\alpha$ = 0.0054 and the final analysis will use a significance level of 0.0492. The interim safety analysis will be performed when 50% of subjects, within their respective cohort, complete their 35 day follow-up. Overall safety will be analyzed first, and if safety outcomes are statistically higher in the treatment group ( $\alpha$ = 0.0054), enrollment will be stopped, participants will be unblinded and each cohort will be analyzed independently. If safety has not been compromised the study maybe resumed after review and recommendation by the SRC. Efficacy will be analyzed for early declaration of success. If power of 90% has been detected and a statistically significant change has been identified ( $\alpha$ = 0.0054), that specific cohort will stop enrollment and the final analysis will be done with completed data from participants enrolled at that time, otherwise the study will continue enrolling patients and final analysis will be completed.

## 10.0 Regulatory, Ethical, and Study Oversight

#### 10.1 Statement of Compliance

This study will be conducted in accordance with this protocol, FDA and applicable local regulatory requirements.

Before enrollment of participants into this study, the IRB will review and approve the protocol, informed consent documents, any promotional material/advertisements, and any other written information to be provided to the participants. The Package Insert for hydroxychloroquine describing the investigational product will be provided to the IRB for review, see Appendix C. Drug information for vitamin D with calcium is provided in Section 6.3. Also see Appendix D. The IRB's composition or a statement that the IRB's composition meets applicable regulatory criteria will be documented.

If the protocol or any other information given to the participant is amended, the revised documents will be reviewed and approved by the IRB, where applicable. The protocol amendment will only be implemented upon the lead site's receipt of approval and, if required, upon the lead site's notification of applicable regulatory authority(ies) approval except for changes necessary to eliminate an immediate hazard to study participants.

#### 10.2 Informed Consent

Written informed consent will embody the elements of informed consent as required by 21 CFR 50.27 and the IRB and will be in accordance with all applicable laws and regulations. Site investigators will enroll participants according to the study eligibility criteria and in compliance with 21 CFR 50, Protection of Human Participants. The investigator will exercise no selectivity so that no bias is introduced from this source.

The site investigator or qualified study team member must obtain documented consent from each potential participant prior to participating in a clinical study or future biomedical research. If there are changes to the participant's status during the study (e.g., health or age of majority requirements), the investigator or study team member delegated this task must ensure the appropriate consent is in place.

A copy of the consent form should be given to the participant before participation in the study.

The initial ICF, any subsequent revised written ICF and any written information provided to the participant must receive Sanford IRB's approval in advance of use. The participant should be informed in a timely manner if new information becomes available that may be relevant to the participant's willingness to continue participation in the study. The communication of this information will be documented in the participant's study chart. Communication may take place in person, over the telephone or by mail.

Specifics about a study and the study population will be added to the consent form template at the protocol level.

#### 10.3 Study Participant Confidentiality

The investigator will comply with applicable participant privacy regulations/guidance as described as per the Health Insurance Portability and Accountability Act (HIPAA) and any additional local regulations.

The lead site is committed to safeguarding participant confidentiality, to the greatest extent possible. Unless required by law, only the investigator, lead site (or representative), IRB, and/or regulatory authorities will have access to confidential medical records that might identify the participant by name.

The participant must be informed that his/her personal study-related data will be used by the lead site in accordance with local data protection law. The level of disclosure must also be explained to the participant.

The participant must be informed that his/her medical records may be examined by Clinical Research Staff for quality data review at each site or other authorized personnel appointed by the lead site, by appropriate IRB members, and by inspectors from regulatory authorities.

#### 10.4 Risks and Benefits

Potential participants will be informed of the risks and benefits of, as well as alternatives to, trial participation. At a minimum, trial designs will take into account the local standard of care.

All participation in clinical trials is voluntary. Participants enter the trial only after informed consent is obtained. Participants may withdraw from a trial at any time, without any influence on their access to, or receipt of, medical care that may otherwise be available to them.

#### 10.5 Ethics

The study protocol, along with the required informed consent forms, will be approved by the Sanford IRB prior to the initiation of any research procedures (at the site). In addition to details described in the sections above (informed consent, confidentiality, and risks and benefits), the investigators should review and consider ethical ramifications in the design and development of this protocol, in accordance with 21 CFR 50. Protections of Human Participants. The investigators will make every effort to minimize and monitor risks and discomforts to participants throughout the course of the study.

#### 10.6 Study Documentation and Case Report Forms (CRFs)

The data collection tool for this study will be defined CRF/eCRFs to be completed by study-site personnel. The investigator will maintain complete and accurate study documentation in a separate file. Study documentation may include medical records/electronic medical records, records detailing the progress of the study for each participant, signed informed consent forms, drug disposition records, correspondence with the IRB and the study monitor/lead site, screening and consent information, CRFs/eCRFs, AE/SAE reports, laboratory reports, participant diaries/questionnaires, data clarifications requested by the lead site study team, and any other documentation

deemed relevant and pertinent to the study and the study participants. Participant data necessary for analysis and reporting will be entered into a validated database or data system in accordance with Title 21 of the Code of Federal Regulations (21 CFR) Part 11. The site investigator is responsible for the procurement of data and for the quality of data recorded on the CRFs/eCRFs.

#### 10.7 Document and Data Retention

Health information will be used to conduct this study to determine research results. Health information is used to report results of research to federal regulatory agencies, if applicable. Health information from study participants may be included in an audit to ensure that the study follows regulations, policies, and study plans.

All records will be maintained indefinitely. Sanford policy on record retention and destruction specific to research studies will be followed for Sanford sites. Non-Sanford sites will follow their policy for record retention and destruction Clinical data will be stored indefinitely. If a subject chooses to withdrawal consent to the study, he/she may request to withdraw. No further data will be collected on the subject, but any data collected prior to withdrawal will be and used for analysis.

The site will retain study documentation and data (electronic case report forms) in accordance with applicable regulatory requirements and each site document and data retention policy.

#### 10.8 Direct Access to Source Data/Documents

The investigator/study site will cooperate and provide direct access to study documents and data, including source documentation for quality data review by the study team at each site, audits by the lead site or lead site's representatives, review by the IRB, and inspections by applicable regulatory authorities. If contacted by an applicable regulatory authority, the investigator will notify the lead site of contact, cooperate with the authority, provide the lead site with copies of all documents received from the authority, and allow the lead site to comment on any responses.

#### 10.9 Protocol Compliance

Deviations from the approved study protocol will be noted by study staff and will be reported to the IRB by the investigator/treating physician per Sanford IRB policy HRP 024 New Information for reporting protocol deviations/violations.

#### **10.10 Publication Policy**

Manuscript submission for publication of the results of this study, or any aspect of work directly related to the study, will be decided by the investigators. Any investigator can submit a publication concept proposal including proposed authorship order to the rest of the investigators for review, which will take place within 30 days after a proposal has been submitted.

## **Appendix A: Abbreviations**

AE / SAE Adverse Event / Serious Adverse Event

BCVA Best Corrected Distance Visual Acuity

CTCAE Common Terminology Criteria for Adverse Events

CDC Center for Disease Control
CFR Code of Federal Regulations
CHF Congestive Heart Failure
CNS Central Nervous System
COVID Coronavirus Disease

**CRF / eCRF** Case Report Form / Electronic Case Report Form

**ECG** Electrocardiogram

**EDC** Electronic Data Capture

**FDA** Food and Drug Administration

GCP Guidelines for Good Clinical Practices

HIPAA Health Insurance Portability and Accountability Act

ICF Informed Consent Form
 IRB Institutional Review Board
 NCI National Cancer Institute
 PI Principal Investigator

**PO** By Mouth

**PPE** Personal Protection Equipment

SARS-CoV-2 Severe acute respiratory syndrome coronavirus 2
SD-OCT Spectral Domain Ocular Coherence Tomography

**SoA** Schedule of Activities

**SOC** Standard of Care

**SRC** Safety Review Committee

VF Visual Field

## **Appendix B: Protocol Amendment History**

| DOCUMENT HISTORY | |
|-------------------|----------------|
| Document | Date |
| [Amendment X] | [Day-Mon-Year] |
| [Amendment X] | [Day-Mon-Year] |
| [Amendment X] | [Day-Mon-Year] |
| Original Protocol | [Day-Mon-Year] |

#### Amendment X

Overall Rationale for the Amendment: (Primary reason for this amendment at the top)

| Section # and<br>Name | Description of Change | Brief Rationale |
|-----------------------|-----------------------|-----------------|
| [INSERT] | [INSERT] | [INSERT] |
| [INSERT] | [INSERT] | [INSERT] |
| [INSERT] | [INSERT] | [INSERT] |

## **Appendix C: Hydroxychloroquine Drug Information**

#### Hydroxychloroquine Sulfate Tablets, USP 200 mg

B. only

DESCRIPTION: Hydroxychioroquine sulfate, USP is a white or practically white, crystalline powder, freely soluble in water; practically insoluble in alcohol, chloroform, and in ether. The chemical name for hydroxychloroquine sulfate is 2-[[4-[(7-Chloro-4-quino)y]amino]pentyl] ethylamino] ethanol sulfate (1:1). Its structural formula is:

The molecular weight of hydroxychiorogulne sulfate is 433.96. and molecular formula is  $C_{18}H_{26}ClN_3O \cdot H_2SO_4$ .

Hydroxychioroquine suitate tablets, USP contain 200 mg hydroxy-

chloroquine sulfate, USP equivalent to 155 mg base, and are for oral

Inactive Ingredients: anhydrous lactose, croscarmellose sodium glyceryl triacetate, hypromellose, magnesium stearate, microcrysta cellulose, polydextrose, polyethylene glycol, povidone, sodium lauryl sulfate and titanium dioxide

CLINICAL PHARMACOLOGY: Pharmacokinetics: Following a single 200 mg oral dose of hydroxychloroquine sulfate tablets to healthy males, the mean peak blood concentration of hydroxychloroquine was 129.6 ng/mL, reached in 3.26 hours with peak concentration was 50.3 ng/ml. reached in 3.74 hours with a half-life of 2963 hours (123.5 days). In the same study, the plasma peak concentration was 50.3 ng/ml. reached in 3.74 hours with a half-life of 2963 hours (123.5 days). Urine hydroxychloroquine levels were still detectable after 3 months with approximately 10% of the dose excreted as the parent drug. Results following a single dose of a 200 mg tablet versus I.v. Infusion (155 mg), demonstrated a half-life of about 40 days and a large volume of distribution. Peak blood concentrations of metabolites were observed at the same time as peak levels of hydroxychloroguine. The mean fraction of united as peak levies of hydroxylinotoquine. The finear inaction of the dose absorbed was 0.74. After administration of single 155 mg and 310 mg intravenous doses, peak blood concentrations ranged from 1161 ng/ml. to 2436 ng/ml. (mean 1918 ng/ml.) following the 155 mg influsion and 6 months following the 310 mg influsion. Pharmacokinetic parameters were not significantly different over the therapeutic dose range of 155 mg and 310 mg indicating linear

Following chronic oral administration of hydroxychloroguine. significant levels of three metabolites, desethylhydroxychioroquine (DHCQ), desethylchioroquine (DCQ), and bidesethylhydroxychioroquine (BDCQ) have been found in plasma and blood, with DHCQ being the major metabolite. The absorption half-life was approximately 3 to 4 hours and the terminal half-life ranged from 40 to 50 days. The long half-life can be attributed to extensive tissue uptake rather than through decreased excretion. Peak plasma levels of hydroxychioroquine were seen in about 3 to 4 hours. Renal clearance in rheumatoid arthritis (RA) patients taking hydroxychloroguine sulfate tablets for at least six months seemed to be similar to that of the single dose studies in volunteers, suggesting that no change occurs with chronic dosing. Range for renal clearance of unchanged drug was approximately 16% to 30% and did not correlate with creatinine clearance; therefore, a dosage adjustment is not required for patients with renal impairment. In RA patients, there was large variability as to the fraction of the dose absorbed (i.e., 30% to 100%), and mean hydroxychioroquine levels were significantly higher in patients with less disease activity. Cellular levels of patients on dally hydroxychlorogulne have been shown to be

hevers of patients of training vigory/introducine and been shown to be higher in mononuclear cells than polymorphonuclear leuccytes. Microbiology: Malaria: Mechanism of Action: The precise mechanism by which hydroxychloroquine exhibits activity against Plasmodium is not known. Hydroxychloroquine, like chloroquine, is a weak base and may exert its effect by concentrating in the acid vesicles of the parasite and by inhibiting polymerization of heme. It can also inhibit certain enzymes by its interaction with DNA.

Activity in vitro and in Clinical Infections: Hydroxychloroquine is active against the erythrocytic forms of chloroquine sensitive strains of Plasmodium faiciparum, Plasmodium malariae, Plasmodium ovale, and Plasmodium vivax. Hydroxychioroquine is not active against the gametocytes and excerythrocytic forms including the hypnozotte stage (P. vivax and P. ovale) of the Plasmodium parasites

Drug Resistance: P. taiciparum strains exhibiting reduced susceptibility to chloroquine also show reduced susceptibility to hydroxychloroquine. Resistance of Plasmodium parasites to chloroquine is widespread (see INDICATIONS AND USAGE: Malarla).

Patients in whom chloroquine or hydroxychloroquine have falled to prevent or cure clinical majaria or parasitemia, or patients who acquired malaria in a geographic area where chloroquine resistance is known to occur should be treated with another form of antimalarial therapy (see INDICATIONS AND USAGE: Maiaria and WARNINGS). Rheumatoid Arthritis and Systemic Lupus Erythematosus: Mechanism of Action: The mechanisms underlying the anti-Inflammatory and Immunomodulatory effects of hydroxychloroquine sulfate tablets are unknown.

INDICATIONS AND USAGE: Malaria: Hydroxychlorogulne sulfate tablets are indicated for the treatment of uncomplicated malaria due to P. faldparum, P. malariae, P. ovale, and P. vivax.

Hydroxychioroquine sulfate tablets are indicated for the prophylaxis of malaria in geographic areas where chloroquine resistance is not

#### Limitations of Use in Malaria:

- Hydroxychloroquine sulfate tablets are not recommended for the treatment of complicated malaria.
- Hydroxychloroquine sulfate tablets are not effective against chloroquine or hydroxychloroquine-resistant strains of Plasmodium species (see CLINICAL PHARMACOLOGY: Microbiology). Hydroxychloroquine sulfate tablets are not recommended for the treatment of malaria acquired in geographic areas where chloroquine resistance occurs or when the *Plasmodium* species has not been identified.

  Hydroxychloroquine sulfate tablets are not recommended for
- malaria prophylaxis in geographic areas where chloroquine resistance occurs.
- Hydroxychioroguine sulfate tablets do not prevent relapses of Priviax or P. ovale because it is not active against the hypno-zofte forms of these parasites. For radical cure of P. vivax and P. ovale infections, concomitant therapy with an 8-aminoquinoline compound is necessary (see CLINICAL PHARMACOLOGY: Microbiology).

Prior to prescribing hydroxychioroquine suifate tablets for the treatment or prophylaxis of malaria, consult the Centers for Disease Control and

Prevention (CDC) Malaria website (http://www.cdc.gov/malaria). **Lupus Erythematosus:** Hydroxychloroquine sulfate tablets are indicated for the treatment of chronic discold lupus erythematosus

and systemic lupus erythematosus in adults.

Rheumatoid Arthritis: Hydroxychloroquine sulfate tablets are Indicated for the treatment of acute and chronic rheumatoid arthritis

CONTRAINDICATIONS: Use of hydroxychioroquine suifate tablets are contraindicated in patients with known hypersensitivity to are contraindicated in patients 4-aminoquinoline compounds.

WARNINGS: Resistant Strains of Malaria: Hydroxychloroquine suifate tablets are not effective against chloroquine-resistant strains of P. faldparum (see CLINICAL PHARMACOLOGY: Microbiology). Ocular: Irreversible retinal damage has been observed in some patients who had received hydroxychlorogulne sulfate. Significant risk factors for retinal damage include daily doses of hydroxychloroquine sultate greater than 6.5 mg/kg (5 mg/kg base) of actual body weight, durations of use greater than five years, subnormal glomerular filtration, use of some concomitant drug products such as tamoxifen citrate and concurrent macular disease.

A baseline ocular examination is recommended within the first year of starting hydroxychioroguine sulfate tablets. The baseline exam should include: best corrected distance visual aculty (BCVA), an automated threshold visual field (VF) of the central 10 degrees (with retesting if an abnormality is noted), and spectral domain ocular coherence tomography (SD-OCT).

For individuals with significant risk factors (daily dose of hydroxychloroquine sulfate greater than 5.0 mg/kg base of actual body weight, subnormal glomerular filtration, use of tamoxifen citrate or concurrent macular disease) monitoring should include annual examinations which include BCVA, VF and SD-OCT. For individuals without significant risk factors, annual exams can usually be deferred until five years of treatment.

In Individuals of Asian descent, retinal toxicity may first be noticed outside the macula. In patients of Asian descent, it is recommended that visual field testing be performed in the central 24 degrees instead of the central 10 degrees

It is recommended that hydroxychloroquine be discontinued if ocular toxicity is suspected and the patient should be closely observed given

that retinal changes (and visual disturbances) may progress even after cessation of therapy.

Cardiac Effects, including Cardiomyopathy and QT Prolongation: Postmarketing cases of life-threatening and fatal cardiomyopathy have been reported with use of hydroxychiorogulne sulfate tablets as well as with use of chloroquine. Patients may present with atrioventricular block, pulmonary hypertension, sick sinus syndrome or with cardiac complications. ECG findings may include atrioventricular, right or left bundle branch block. Signs or symptoms of cardiac compromise have appeared during acute and chronic treatment. Clinical monitoring for signs and symptoms of cardiomyopathy is advised, including use of appropriate diagnostic tools such as ECG to monitor patients for cardiomyopathy during hydroxychioroquine sulfate tablets therapy. Chronic toxicity should be considered when conduction disorders (bundle branch block/atrio-ventricular heart block) or biventricular hypertrophy are diagnosed. If cardiotoxicity is suspected, prompt discontinuation of hydroxychlorogulne sulfate tablets may prevent life-threatening complications.

Hydroxychloroquine sulfate tablets prolong the QT Interval. Ventricular arrhythmias and torsades de pointes have been reported in patients taking hydroxychloroquine sulfate tablets (see OVERDOSAGE). Therefore, hydroxychloroquine suifate tablets should not be administered with other drugs that have the potential to prolong the QT interval (see DRUG INTERACTIONS).

Worsening of Psoriasis and Porphyria: Use of hydroxychioroquine sulfate tablets in patients with psoriasis may precipitate a severe attack of psoriasis. When used in patients with porphyria the condition may be exacerbated. The preparation should not be used in these conditions unless in the judgment of the physician the benefit to the patient outweighs the possible hazard.

Proximal Myopathy and Neuropathy: Skeletal muscle myopathy or neuropathy leading to progressive weakness and atrophy of proximal muscle groups, depressed tendon reflexes, and abnormal nerve conduction, have been reported. Muscle and nerve blopsles have been associated with curvilinear bodies and muscle fiber atrophy with vacuolar changes. Assess muscle strength and deep tendon reflexes periodically in patients on long-term therapy with hydroxychloroguine sulfate tablets.

Neuropsychiatric Events, including Suicidality: Suicidal behavior has been rarely reported in patients treated with hydroxychloroguine sulfate tablets

Hypoglycemia: Hydroxychloroguine sulfate tablets have been shown to cause severe hypoglycemia including loss of consciousness that could be life-threatening in patients treated with or without antidiabetic medications (see DRUG INTERACTIONS and ADVERSE REACTIONS). Patients treated with hydroxychloroquine sulfate tablets should be warned about the risk of hypoglycemia and the associated clinical signs and symptoms. Patients presenting with clinical symptoms suggestive of hypoglycemia during treatment with hydroxychioroquine suitate tablets should have their blood glucose checked and treatment reviewed as

PRECAUTIONS: General: Use with caution in patients with gastrointestinal, neurological, or blood disorders, and in those with a sensitivity to quinine.

Hepactic/Renal Disease: Antimalarial compounds should be used with caution in patients with hepatic disease or alcoholism or in conjunction with known hepatotoxic drugs. A reduction in dosage may be necessary in patients with hepatic or renal disease, as well as in those taking medicines known to affect these organs.

Hematologic Effects/Laboratory Tests: Antimalarial compounds should be used with caution in patients with hepatic disease or alcoholism or in conjunction with known hepatotoxic drugs.

Periodic blood cell counts should be performed if patients are given prolonged therapy. If any severe blood disorder such as aplastic anemia, agranulocytosis, leukopenia, or thrombocytopenia, appears which is not attributable to the disease under treatment, consider

discontinuation of hydroxychioroquine sulfate tablets.
Hydroxychioroquine sulfate tablets should be administered with caution in patients having glucose-6-phosphate dehydrogenase (G-6-PD) deficiency.

Dermatologic Effects: Dermatologic reactions to hydroxychloroquine sulfate tablets may occur and, therefore, proper care should be exercised when it is administered to any patient receiving a drug with

a significant tendency to produce dematitis.

Drug Interactions: Digoxin: Concomitant hydroxychloroquine suitate tablets and digoxin therapy may result in increased serum digoxin levels: serum digoxin levels should be closely monitored in patients receiving combined therapy.

Insulin or Antidiabetic Drugs: As hydroxychioroquine suifate tablets may enhance the effects of a hypoglycemic treatment, a decrease in doses of insulin or antidiabetic drugs may be required.

#### Protocol PEPCOH

Drugs that Prolong QT Interval and Other Arrhythmogenic Drugs: Drugs that Proong of interval and other Armynmogenic brugs: Hydroxychioroguline sulfate tablets prolong the OT interval and should not be administered with other drugs that have the potential to induce cardiac armyfhmias. Also, there may be an increased risk of inducing ventricular armyfhmias if hydroxychioroquine sulfate tablets are used concomitantly with other armyfhmogenic drugs.

Mefloquine and Other Drugs Known to Lower the Convulsive Threshold: Hydroxychloroquine sulfate tablets can lower the convulsive threshold. Co-administration of hydroxychloroquine sulfate tablets with other antimalariais known to lower the convulsion threshold (e.g., mefloguine) may increase the risk of convulsions.

Antiepileptics: The activity of antiepileptic drugs might be impaired if co-administered with hydroxychioroquine sulfate tablets.

Methotrexate: Combined use of methotrexate with hydroxychioroquine

sulfate tablets have not been studied and may increase the incidence of adverse effects

Cyclosporin: An increased plasma cyclosporin level was reported when cyclosporin and hydroxychloroquine sulfate tablets were co-administered

The following interactions have been observed on treatment with the structurally related substance chloroquine phosphate, and therefore cannot be ruled out for hydroxychloroquine.

Praziquantel: Chloroquine has been reported to reduce the bloavailability of praziquantel.

Antacids and Kaolin: Antacids and kaolin can reduce absorption of

chloroquine; an interval of at least 4 hours between intake of these agents and chloroguine should be observed.

Cimetidine: Cimetidine can inhibit the metabolism of chloroquine, increasing its plasma level. Concomitant use of cimetidine should be avoided.

Ampicilin: In a study of healthy volunteers, chloroquine significantly reduced the bloavailability of ampicillin.

Information for Patients: Patients should be informed of the early

signs and symptoms of toxicity such as rash or visual changes. Patients must see their physicians promptly in case of the appearance of these or of any unusual effects. Perfodic laboratory tests may be recommended in some patients. Patients should be fully informed of the potential risks of the use of hydroxychloroquine sulfate tablets, especially in pregnancy and in children.

Carcinogenesis, Mutagenesis, Impairment of Fertility: Long-term studies in animals have not been conducted to evaluate the carcinogenic potential of hydroxychloroquine sulfate tablets.

The mutagenic potential of hydroxychloroquine was not evaluated, owever, chloroquine has been shown to be a catalytic inhibitor of DNA repair enzymes (topolsomerase II) and to produce weak genotoxic effects through this mode of action.

Pregnancy: Teratogenic Effects: Human pregnancies resulting in live births have been reported in the literature and no increase in the rate of birth defects has been demonstrated. Embryonic deaths and malformations of anophthalmia and microphthalmia in the offspring have been reported when pregnant rats received large doses of chlorogulne.

Nursing Mothers: Caution should be exercised when administering hydroxychioroquine sulfate tablets to nursing women. It has been demonstrated that hydroxychioroquine administered to nursing women is excreted in human milk and it is known that intants are extremely sensitive to the toxic effects of 4-aminoquinolines.

Pediatric Use: Safely and efficacy have not been established in the chronic use of hydroxychloroquine sulfate tablets for systemic lupus erythematosus and juvenile idiopathic arthritts in children. Children are especially sensitive to the 4-aminoquinoline compounds. Most reported fatalities followed the accidental indestion of chloroguine. sometimes in small doses (0.75 g or 1 g in one 3-year-old child). Patients should be strongly warned to keep these drugs out of the reach of children (see OVERDOSAGE).

Geriatric Use: Clinical studies of hydroxychloroguine sulfate tablets Genatic user: Climical studies on injurioxyclimicordurine suriate italies did not include sufficient numbers of subjects aged 65 and over to determine whether they respond differently from younger subjects. However, this drug is known to be substantially excreted by the kidney, and the fisk of toxic reactions to this drug may be greater in patients with impaired renal function. Because elderly patients are more likely to have decreased renal function, care should be taken in dose selection and it may be useful to monitor renal function.

ADVERSE REACTIONS: The following adverse reactions have been identified during post-approval use of hydroxychioroquine sulfate labiets or other 4-aminoqunoline compounds. Because these reactions are reported voluntarily from a population of uncertain size, it is not always possible to reliably estimate their frequency or establish a causal relationship to drug exposure

Blood and Lymphatic System Disorders: Bone marrow fallure, anemia, aplastic anemia, agranulocytosis, leukopenia, and

thrombocytopenia. Hemolysis reported in Individuals with glucose-6phosphate dehydrogenase (G-6-PD) deficiency

Cardiac Disorders: Cardiomyopathy which may result in cardiac failure and in some cases a fatal outcome (see WARNINGS and OVERDOSAGE). Hydroxychloroquine sulfate tablets prolong the QT Interval. Ventricular arrhythmias and torsade de pointes have been reported in patients taking hydroxychioroguine sulfate tablets (see OVERDOSAGE and DRUG INTERACTIONS).

Ear and Labyrinth Disorders: Vertigo, tinnitus, nystagmus, nerve deafness, deafness.

Eye Disorders: Irreversible retinopathy with retinal pigmentation changes (bull's eye appearance), visual field defects (paracentral scotomas) and visual disturbances (visual acuity, maculopathies (macular degeneration), decreased dark adaptation, color vision abnormalities, corneal changes (edema and opacities) including comeal deposition of drug with or without accompanyling symptoms (halo around lights, photophobia, blurred vision).

Gastrointestinal Disorders: Nausea, vomitling, diarrhea, and

abdominal pain.

General Disorders and Administration Site Conditions: Fatique Hepatobiliary Disorders: Liver function tests abnormal, hepatic

Immune System Disorders; Urticaria, angloedema, bronchospasm. Metabolism and Nutrition Disorders: Decreased appetite, hypoglycemia, porphyria, weight decreased.

Musculoskeletal and Connective Tissue Disorders: Sensorimotor disorder, skeletal muscle myopathy or neuromyopathy leading to progressive weakness and atrophy of proximal muscle groups, depression of tendon reflexes and abnormal nerve conduction.

Nervous System Disorders: Headache, dizziness, seizure, ataxia and extrapyramidal disorders such as dystonia, dyskinesia, and tremor have been reported with this class of drugs.

Psychiatric Disorders: Affect/emotional lability, nervousness,

irritability, nightmares, psychosis, suicidal behavior.

Skin and Subcutaneous Tissue Disorders: Rash, pruritus, pigmentation disorders in skin and mucous membranes, hair color changes, alopecia. Dermatitis bullous eruptions including erythema multiforme, Stevens-Johnson Syndrome, and toxic epidermal necrolysis, drug reaction with eosinophilia and systemic symptoms (DRESS syndrome), photosensitivity, dematitis exfoliative, acute generalized exanthematous pustulosis (GREP). AGEP has to be distinguished from psoffasis, although hydroxychioroquine suitate tablets may precipitate attacks of psoriasis. It may be associated with pyrexia and hyperleukocytosis.

To report SUSPECTED ADVERSE REACTIONS, contact Mylan Pharmaceuticals Inc. at 1-877-446-3679 (1-877-4-INFO-RX) or FDA at 1-800-FDA-1088 or www.fda.gov/medwatch.

OVERDOSAGE: The 4-aminoquinoline compounds are very rapidly and completely absorbed after ingestion, and in accidental overdosage, or rarely with lower doses in hypersensitive patients, toxic symptoms may occur within 30 minutes. The symptoms of overdosage may include headache, drowsiness, visual disturbances, cardiovascular collapse, convulsions, hypokalemial, rhythm and conduction disorders including QT prolongation, torsades de pointes, ventricular tachycardia and ventricular fibrillation, followed by sudden potentially fatal respiratory and cardiac arrest. Treatment is symptomatic and must be prompt. Immediate gastric lavage until the stomach is completely emptied is indicated. After lavage, activated charcoal is introduced by the stomach tube within 30 minutes of ingestion of the drug may inhibit further intestinal absorption. To be effective, the dose of activated charcoal should be at least flux times the activated dose. activated charcoal should be at least five times the estimated dose of

hydroxychioroquine ingested.

Consideration should be given to administering diazepam parenterally since studies suggest that it may be beneficial in reversing chlorogulne and hydroxychlorogulne cardiotoxicity.

Respiratory support and shock management should be instituted as necessary.

Exchange transfusions are used to reduce the level of 4-aminoquinoline drug in the blood.

A patient who survives the acute phase and is asymptomatic should be closely observed for at least six hours. Fluids may be forced and sufficient ammonlum chloride (8 g dally in divided doses for adults) may be administered for a few days to acidify the urine. This will promote urinary excretion in cases of both overdosage and sensitivity. However, caution must be exercised in patients with impaired renal function and/or metabolic acidosis.

DOSAGE AND ADMINISTRATION: One hydroxychloroquine sulfate tablet contains 200 mg of hydroxychloróquiné sulfaté, which is equivalent to 155 mg base

Take hydroxychlorogulne sulfate tablets with a meal or a glass

of milk

Malaria: Prophylaxis: Adults: 400 mg (310 mg base) once weekly on the same day of each week starting 2 weeks prior to exposure, and continued for 4 weeks after leaving the endemic area.

and continued for 4 weeks after leaving the endemic area. Weight-Based Doshig in Adults and Podelatic Patients: 6.5 mg/kg (5 mg/kg base), not to exceed 400 mg (310 mg base), once weekly on the same day of the week starting 2 weeks prior to exposure, and continued for 4 weeks after leaving the endemic area. Treatment of Uncomplicated Malaria: Adults: 800 mg (620 mg base) followed by 400 mg (310 mg base) at 6 hours, 24 hours and 48 hours after the Initial dose (total 2000 mg hydroxychioroquine sulfate or 1550 mg base).

Weight Based Dosage in Adults and Pediatric Patients: 13 mg/kg Weight based busage in Adults and Pedaritis Tallents: 1 tillying (10 mg/kg base), not to exceed 800 mg (620 mg base); followed by 6.5 mg/kg (5 mg/kg base), not to exceed 400 mg (310 mg base), at 6 hours, 24 hours and 48 hours after the Initial dose, Hydroxychloroquine sulfate tablets film-coated tablets cannot be divided, therefore they should not be used to treat patients who weigh less than 31 kg.

For radical cure of P. vivax and P. malariae infections, concomitant

therapy with an 8-aminoquinoline compound is necessary. **Lupus Erythematosus:** The recommended adult dosage is 200 mg to 400 mg (155 mg to 310 mg base) dally, administered as a single dally dose or in two divided doses. Doses above 400 mg a day are not recommended.

The incidence of retinopathy has been reported to be higher when this maintenance dose is exceeded.

Rheumatold Arthritis: The action of hydroxychloroquine is cumulative and may require weeks to months to achieve the maximum therapeutic effect (see CLINICAL PHARMACOLOGY).

Initial Adult Dosage: 400 mg to 600 mg (310 mg to 465 mg base) dally, administered as a single dally dose or in two divided doses. In

a small percentage of patients, side effects may require temporary reduction of the initial dosage. Maintenance Adult Dosage: When a good response is obtained, the dosage may be reduced by 50 percent and continued at a maintenance level of 200 mg to 400 mg (155 mg to 310 mg base) daily, administered as a single daily dose or in two divided doses.

Do not exceed 600 mg or 6.5 mg/kg (5 mg/kg base) per day, whichever is lower, as the incidence of retinopathy has been reported to be higher when this maintenance dose is exceeded.

Corticosteroids and salicylates may be used in conjunction with hydroxychioroquine sulfate tablets, and they can generally be decreased gradually in dosage or eliminated after a maintenance dose of hydroxychioroquine sulfate tablets has been achieved.

HOW SUPPLIED: Hydroxychloroquine Sulfate Tablets, USP are available containing 200 mg of hydroxychloroquine sulfate, USP, equivalent to 155 mg of base.

The 200 mg tablets are white, film-coated, round, unscored tablets debossed with M on one side of the tablet and 373 on the other side. They are available as follows:

NDC 0378-0373-01

Store at 20° to 25°C (68° to 77°F). [See USP Controlled Room Temperature.]

Dispense in a tight, light-resistant container as defined in the USP

using a child resistant closure. Keep out of the reach of children.

Do not crush or divide hydroxychloroquine sulfate film-coated tablets (see DOSAGE AND ADMINISTRATION).



Mylan Pharmaceuticals Inc. Morgantown, WV 26505 U.S.A.

HXCQ:R10

## **Appendix D: Exclusion Medication List**

| Digoxin | Praziquantel |
|--------------------|------------------------|
| Mefloquine | Antacids |
| Tamoxifen citrate | Kaolin |
| Methotrexate | Cimetidine |
| Cyclosporine | Ampicillin |
| Insulin | Laxatives |
| Antidiabetic drugs | Enemas |
| Loop diuretics | Amphotericin B |
| Thiazides | High dose |
| | corticosteroids |
| Pyridostigmine | Proton pump inhibitors |
| | Neostigmine |
| | Pyridostigmine |

## CredibleMeds Filtered QTDrug List



The last revision date: March 19, 2020

See Note below for safe use of this Table

The drug list below contains drugs from the categories: Known Risk of TdP, Possible

Risk of TdP AND filtered by

Market filter: Only Drugs on US Market AND filtered by Keyword --> " "

| Generic<br>Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Alfuzosin | Uroxatral | Alpha-1 adrenergic blocker | Benign<br>prostatic<br>hyperplasia | Possible Risk of TdPAnd Avoid in congenital long QT | oral |
| Amiodarone | Cordarone, Pacerone, Nexterone | Antiarrhythmic | Arrhythmia | Risk of TdPAnd Avoid in congenital long QT | oral,<br>injectio<br>n |
| Anagrelide | Agrylin, Xagrid | Phosphodiesterase 3 inhibitor | Thrombocythe mia | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral |
| Apalutamide | Erleada | Nonsteroidal<br>antiandrogen | Cancer<br>(prostate) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Apomorphine | Apokyn, Ixense,<br>Spontane, Uprima | Dopamine agonist | Parkinson's<br>disease | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>sublingua<br>I,<br>injection |
| Aripiprazole | Abilify, Aripiprex | Antipsychotic,<br>atypical | Schizophrenia,<br>depression<br>(adjunct) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injectio<br>n |
| Arsenic trioxide | Trisenox | Anti-cancer | Cancer<br>(leukemia) | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | injection |

#### CONFIDENTIAL

#### Protocol PEPCOH

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Artemether/Lumefantrin e | Coartem | Anti-malarial | Marlaria | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Asenapine | Saphris, Sycrest | Antipsychotic,<br>atypical | Schizophrenia | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | sublingual |
| Atomoxetine | Strattera | CNS stimulant | ADHD | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Azithromycin | Zithromax, Zmax | Antibiotic | Bacterial infection | Risk of TdPAnd Avoid in congenital long QT | oral,<br>injection |
| Bedaquiline | Sirturo | Antibiotic | Tuberculosis,<br>Multi-drug<br>resistant | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Bendamustine | Treanda, Treakisym,<br>Ribomustin, Levact | Anti-cancer | Cancer<br>(Leukemia,<br>lymphoma) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Bepridil | Vascor | Antianginal | Angina Pectoris<br>(heart pain) | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral |
| Betrixaban | Веvухха | Anticoagulant | Anticoagulant | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Bortezomib | Velcade, Bortecad | Proteasome inhibitor | Cancer (multiple<br>myeloma,<br>lymphoma) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Bosutinib | Bosulif | Anti-cancer | Cancer (leukemia) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Buprenorphine | Butrans, Belbuca, Bunavail,<br>Buprenex, Subutex,<br>Suboxone, Zubsolv | Opioid agonist | Narcotic<br>addiction and<br>pain | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | sublingual,<br>topical,<br>injection |
| Cabozantinib | Cometriq | Anti-cancer | Cancer (renal cell) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Capecitabine | Xeloda | Anti-cancer | Cancer (GI,<br>Breast) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Ceritinib | Zykadia | Anti-cancer | Cancer (Lung) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Cesium Chloride | Energy Catalyst | Toxin | Alternative<br>therapy<br>cancer | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Chloroquine | Aralen | Antimalarial | Malaria | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Chlorpromazine | Thorazine, Largactil,<br>Megaphen | Antipsychotic /<br>Antiemetic | Nausea,<br>Schizophrenia,<br>many others | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral,<br>injection,<br>suppository |
| Cilostazol | Pletal | Phosphodiesterase 3 inhibitor | Intermittental | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Ciprofloxacin | Cipro, Cipro-XR, Neofloxin | Antibiotic | Bacterial<br>infection | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Citalopram | Celexa, Cipramil | Antidepressant,<br>SSRI | Depression | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Clarithromycin | Biaxin, Prevpac | Antibiotic | Bacterial infection | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral,<br>inhaled |
| Clozapine | Clozaril, Fazaclo, Versacloz | Antipsychotic,<br>atypical | Schizophrenia | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Cobimetinib | Cotellic | Anti-cancer | Cancer<br>(Melanoma) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Crizotinib | Xalkori | Anti-cancer | Cancer (Non-<br>small cell lung<br>cancer,<br>metastatic) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Dabrafenib | Tafinlar | Anti-cancer | Cancer<br>(melanoma) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Dasatinib | Sprycel | Anti-cancer | Cancer (leukemia) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Degarelix | Firmagon, Ferring | Anti-androgen | Cancer (prostate) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection,<br>suppository |
| Desipramine | Pertofrane, Norpramine | Antidepressant,<br>Tricyclic | Depression | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Deutetrabenazine | Austedo | Vesicular monamine transporter 2 inhibitor | Chorea<br>(Huntington's<br>disease) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |

| Conorio Namo | Brand Names (Partial List) | Drug Class | Thereneutic Hee | Diek Catagony | Doute |
|---|---|---|---|---|---|
| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic Use | Risk Category | Route |
| Dextromethorphan/Quini | Nuedexta | Unknown | Pseudobulbar affect | Possible Risk | oral |
| dine | | | | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Disopyramide | Norpace | Antiarrhythmic | Arrhythmia | Risk of | oral, |
| | | | | TdPAnd | injection |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Dofetilide | Tikosyn | Antiarrhythmic | Arrhythmia | Risk of | oral |
| | | | | TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Dolasetron | Anzemet | Antiemetic | Nausea, vomiting | Possible Risk | oral, |
| | | | | of TdPAnd | injection |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Donepezil | Aricept | Cholinesterase | Dementia (Alzheimer's | Risk of | oral |
| | | inhibitor | Disease) | TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Dronedarone | Multaq | Antiarrhythmic | Arrhythmia | Risk of | oral |
| | | | | TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Efavirenz | Sustiva | Antiviral | HIV/AIDS | Possible Risk | oral |
| | | | | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Eliglustat | Cerdelga | Glucosylceramide | Gaucher's disease | Possible Risk | oral |
| | | synthase inhibitor | | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| | | | I | 3, - | |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Encorafenib | Braftovi | BRAF inhibitor | Cancer<br>(Melanoma) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Entrectinib | Rozlytrek | Anti-cancer | Cancer (Lung) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Epirubicin | Ellence, Pharmorubicin,<br>Epirubicin Ebewe | Anti-cancer | Cancer | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Eribulin mesylate | Halaven | Anti-cancer | Cancer (breast, metastatic) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Erythromycin | E.E.S., Robimycin, EMycin, Erymax, Ery-Tab, Eryc Ranbaxy, Erypar, Eryped, Erythrocin Stearate Filmtab, Erythrocot, E-Base, Erythroped, Ilosone, MY-E, Pediamycin, Abboticin, Abboticin-ES, Erycin, PCE Dispertab, Stiemycine, Acnasol, Tiloryth | Antibiotic | Bacterial<br>infection,<br>increase GI<br>motility | Risk of TdPAnd<br>Avoid in<br>congenital long<br>QT | oral,<br>injection |
| Escitalopram | Cipralex, Lexapro, Nexito, Anxiset-E, Exodus, Esto, Seroplex, Elicea, Lexamil, Lexam, Entact, Losita, Reposil, Animaxen, Esitalo, Lexamil | Antidepressant,<br>SSRI | Depression<br>(major),<br>anxiety<br>disorders | Risk of TdPAnd<br>Avoid in<br>congenital long<br>QT | oral |
| Ezogabine (Retigabine) | Potiga, Trobalt | Anticonvulsant | Seizures, Partial | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Felbamate | Felbatol | Anticonvulsant | Seizures | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |

| | 1100001 | | | | |
|---|---|---|---|---|---|
| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
| Fingolimod | Gilenya | Sphingosine phospate receptor modulator | Multiple Sclerosis | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Flecainide | Tambocor, Almarytm,<br>Apocard, Ecrinal, Flécaine | Antiarrhythmic | Arrhythmia | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral |
| Fluconazole | Diflucan, Trican | Antifungal | Fungal infection | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral,<br>injection |
| Fluorouracil (5-FU) | Adrucil, Carac, Efudex,<br>Efudix | Anti-cancer | Cancer | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Gemifloxacin | Factive | Antibiotic | Bacterial infection | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Gilteritinib | Xospata | Antineoplastic | Cancer (Acute<br>Myeloid<br>Leukemia) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Glasdegib | Daurismo | Anti-cancer | Cancer (Acute<br>myeloid leukemia) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Granisetron | Kytril, Sancuso, Granisol | Antiemetic | Nausea, vomiting | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection,<br>topical |
| Haloperidol | Haldol, Aloperidin, Bioperidolo, Brotopon, Dozic, Duraperidol, Einalon S, Eukystol, Halosten, Keselan, Linton, Peluces, Serenace, Serenase, Sigaperidol | Antipsychotic | Schizophrenia, agitation | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral,<br>injection |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic Use | Risk Category | Route |
|---|---|---|---|---|---|
| Hydrocodone - ER | Hysingla™ ER, Zohydro ER | Analgesic | Pain, severe | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>suppository |
| Hydroxychloroquine | Plaquenil, Quineprox | Antimalarial,<br>Anti-inflammatory | Malaria, SLE,<br>rheumatoid<br>arthritis | Risk of TdPAnd Avoid in congenital long QT | oral |
| lloperidone | Fanapt, Fanapta, Zomaril | Antipsychotic,<br>atypical | Schizophrenia | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Imipramine<br>(Melipramine) | Tofranil | Antidepressant,<br>Tricyclic | Depression | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Inotuzumab ozogamicin | Besponsa | Anti-cancer | Cancer (acute<br>lymphocytic<br>leukemia} | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Isradipine | Dynacirc | Antihypertensive | Hypertension | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Ivosidenib | Tibsovo | IDH1 inhibitor | Cancer (Acute<br>myeloid leukemia) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Lapatinib | Tykerb, Tyverb | Anti-cancer | Cancer (breast, metastatic) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Lefamulin | Xenleta | Antibiotic | Community<br>acquired<br>pneumonia | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Lenvatinib | Lenvima | Anti-cancer | Cancer (Thyroid) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Leuprolide (Leuprorelin) | Lupron, Eligard, Viadur,<br>Carcinil, Enanton, Leuplin,<br>Lucrin, Procren, Prostap | Anti-androgen | Cancer (prostate) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Levofloxacin | Levaquin, Tavanic | Antibiotic | Bacterial infection | Risk of TdPAnd Avoid in congenital long QT | oral,<br>injection |
| Lithium | Eskalith, Lithobid | Antimanic | Bipolar disorder | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Lofexidine | Lucemyra | Alpha-2-adrenergic agonist, central | Opioid<br>withdrawal<br>syndrome | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Lopinavir/Ritonavir | Kaletra, Aluvia | Antiviral | HIV/AIDS | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Lumateperone | Caplyta | Antipsychotic,<br>atypical | Schizophrenia | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Lurasidone | Latuda | Antipsychotic,<br>atypical | Schizophrenia,<br>biopolar disorder<br>and others | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Maprotiline | Ludiomil | Anti-depressant,<br>Tetracyclic | Depression | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Memantine | Namenda XR | NMDA receptor antagonist | Alzheimer's<br>disease | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Methadone | Dolophine, Symoron,<br>Amidone, Methadose,<br>Physeptone, Heptadon | Opioid agonist | Narcotic<br>dependence,<br>pain | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral,<br>injection |
| Midostaurin | Rydapt | Anti-cancer | Cancer<br>(Acute<br>myeloid<br>leukemia) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Mifepristone | Korlym, Mifeprex | Progesterone antagonist | Pregnancy<br>termination | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Mirabegron | Myrbetriq | Beta3 adrenergic antagonist | Bladder spasm | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Mirtazapine | Remeron | Antidepressant,<br>Tetracyclic | Depression | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Moexipril/Hydrochlorothi azide | Uniretic, Univasc | Antihypertensive | Hypertension, diuresis | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Moxifloxacin | Avelox, Avalox, Avelon | Antibiotic | Bacterial infection | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral,<br>injection |
| Necitumumab | Portrazza | Anti-cancer | Cancer (Lung) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Nicardipine | Cardene | Antihypertensive | Hypertension | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Nilotinib | Tasigna | Anti-cancer | Cancer (leukemia) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |

| | 1.0000 | TTET COTT | | | |
|---|---|---|---|---|---|
| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
| Nortriptyline | Pamelor, Sensoval, Aventyl,<br>Norpress, Allegron, Noritren,<br>Nortrilen | Antidepressant,<br>Tricyclic | Depression | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Nusinersen | Spinraza | Antisense oligonucleotide | Spinal Muscular<br>Atrophy | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Ofloxacin | Floxin | Antibiotic | Bacterial infection | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Ondansetron | Zofran, Anset, Ondemet,<br>Zuplenz, Emetron, Ondavell,<br>Emeset, Ondisolv, Setronax | Antiemetic | Nausea, vomiting | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral,<br>injection,<br>suppository |
| Osimertinib | Tagrisso | Anti-cancer | Cancer (EGFR pos. NSC Lung cancer) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Oxaliplatin | Eloxatin | Anti-cancer | Cancer | Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | injection |
| Paliperidone | Invega, Xepilon | Antipsychotic,<br>atypical | Schizophrenia | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Palonosetron | Aloxi | Antiemetic | Nausea, vomiting | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Panobinostat | Farydak | Histone deacetylase inhibitor | Cancer, Multiple<br>myeloma | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic Use | Risk Category | Route |
|---|---|---|---|---|---|
| Pasireotide | Signifor | Somatostatin analog | Cushings Disease | Possible Risk<br>of TdPAnd<br>Avoid in | injection,<br>topical |
| | | | | congenital<br>long QT | |
| Pazopanib | Votrient | Anti-cancer | Cancer (renal cell, sarcoma) | Possible Risk<br>of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Pentamidine | Pentam | Antifungal | Fungal infection<br>(Pneumocystis<br>pneumonia) | Risk of<br>TdPAnd<br>Avoid in<br>congenital<br>long QT | injection,<br>inhaled |
| Perphenazine | Trilafon, Etrafon/Triavil, Decentan | Antipsychotic | Schizophrenia | Possible Risk<br>of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Pimavanserin | Nuplazid | Antipsychotic,<br>atypical | Psychosis,<br>Parkinson's Disease | Possible Risk<br>of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Pimozide | Orap | Antipsychotic | Tourette's Disorder | Risk of<br>TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Pitolisant (Tiprolisant) | Wakix | Histamine 3<br>antagonist/inverse<br>agonist | Narcolepsy | Possible Risk<br>of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Pretomanid | | Antitubercular | Tuberculosis,<br>extensively drug<br>resistant | Possible Risk<br>of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |

| | | T El COIT | | | |
|---|---|---|---|---|---|
| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic Use | Risk Category | Route |
| Primaquine phosphate | | Antimalarial | Malaria | Possible Risk | oral |
| | | | | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Procainamide | Pronestyl, Procan | Antiarrhythmic | Arrhythmia | Risk of | injection |
| | | | | TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Promethazine | Phenergan | Antipsychotic / | Nausea, vomiting | Possible Risk | oral, |
| | | Antiemetic | | of TdPAnd | injection, |
| | | | | Avoid in | suppository |
| | | | | congenital | |
| | | | | long QT | |
| Quinidine | Quinaglute, Duraquin, | Antiarrhythmic | Arrhythmia | Risk of | oral, |
| | Quinact, Quinidex, Cin-Quin, | | | TdPAnd | injection |
| | Quinora | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Ribociclib | Kisqali | Anti-cancer | Cancer (breast) | Possible Risk | oral |
| | | | | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Rilpivirine | Edurant, Complera, Eviplera, | Antiviral | Viral infection | Possible Risk | oral |
| | Juluca | | (HIV/AIDS) | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Romidepsin | Istodax | Histone deacetylase | Cancer (lymphoma) | Possible Risk | injection |
| | | inhibitor | | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |
| Saquinavir | Invirase(combo) | Antiviral | Viral infection | Possible Risk | oral |
| | | | (HIV/AIDS) | of TdPAnd | |
| | | | | Avoid in | |
| | | | | congenital | |
| | | | | long QT | |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Siponimod | Mayzent | | Multiple Sclerosis | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Sorafenib | Nexavar | Anti-cancer | Cancer (liver,<br>renal cell,<br>metastatic<br>thyroid) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Sotalol | Betapace, Sotalex, Sotacor | Antiarrhythmic | Arrhythmia | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Sunitinib | Sutent | Anti-cancer | Cancer (GIST,<br>renal cell,<br>pNET) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Tacrolimus | Prograf, Prograf, Advagraf,<br>Protopic | Immunosuppressant | Immune<br>suppression | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Tamoxifen | Nolvadex, Istubal | Anti-cancer | Cancer (breast) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Tazemetostat | Tazverik | Anti-cancer | Epithelioid<br>sarcoma | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Telavancin | Vibativ | Antibiotic | Bacterial infection | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | injection |
| Tetrabenazine | Nitoman, Xenazine | Vesicular Monoamine Transporter 2 Inhibitor | Chorea<br>(Huntington's<br>disease) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |

| Generic Name | Brand Names (Partial List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Thioridazine | Mellaril, Novoridazine, Thioril | Antipsychotic | Schizophrenia | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Tipiracil/Trifluridine | Lonsurf | Anti-cancer | Cancer<br>(Metastatic<br>colorectal) | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Tizanidine | Zanaflex, Sirdalud | Muscle relaxant | Muscle<br>spasticity | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Tolterodine Toremifene | Detrol, Detrusitol | Muscle relaxant | Bladder spasm | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT<br>Possible Risk of | oral |
| Toremilene | Fareston | Estrogen agonist/antagonist | Cancer (breast, metastatic) | TdPAnd Avoid in congenital long QT | oral |
| Tramadol | Crispin, Ralivia ER, Ralivia<br>Flashtab, Tramadolum,<br>Tramal, Tramodol, Tridural,<br>Ultram, Ultram ER, Zydol,<br>Ixprim, Zaldiar, Topalgic | Analgesic | Pain | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection,<br>suppository |
| Trimipramine | Surmontil, Rhotrimine,<br>Stangyl | Antidepressant,<br>Tricyclic | Depression | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |
| Valbenazine | Ingrezza | Vesicular monamine<br>transporter 2 inhibitor | Tardive<br>Dyskinesia | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral |
| Vandetanib | Caprelsa | Anti-cancer | Cancer (thyroid) | Risk of TdPAnd<br>Avoid in<br>congenital<br>long QT | oral |
| Vardenafil | Levitra | Phosphodiesterase 5 inhibitor | Erectile<br>dysfunction | Possible Risk of<br>TdPAnd Avoid in<br>congenital<br>long QT | oral,<br>injection |

| Generic Name | Brand Names (Partial<br>List) | Drug Class | Therapeutic<br>Use | Risk Category | Route |
|---|---|---|---|---|---|
| Vemurafenib | Zelboraf | Anti-cancer | Cancer<br>(melanoma) | Possible Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral |
| Venlafaxine | Effexor, Efexor | Antidepressant,<br>SNRI | Depression | Possible Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral |
| Vorinostat | Zolinza | Histone deacetylase inhibitor | Cancer<br>(lymphoma) | Possible Risk of<br>TdPAnd Avoid<br>in congenital<br>long QT | oral |

Note: Medicines on this list are reviewed on an ongoing basis to assure that the available evidence supports their continued placement on this list. The list changes regularly and we recommend checking the website at crediblemeds.org for the most up-to-date information. There may be many additional brand names that are not listed on this form.

Disclaimer and Waiver: The information presented is intended solely for the purpose of providing general information about

health-related matters. It is not intended for any other purpose, including but not limited to medical advice and/or treatment, nor is it intended to substitute for the users' relationships with their own health care providers. To that extent, by use of this website and the information it contains, the user affirms the understanding of the purpose and releases AZCERT, Inc. from any claims arising out of his/her use of the website and its lists. The absence of drugs from these lists should not be considered an indication that they are free of risk of QT prolongation or torsades de pointes. Many medicines have not been tested for this risk in patients, especially those with congenital long QT syndrome.

# **Appendix E: References**

Haeusler IL, Chan XHS, Guerin PJ, White NJ. The arrhythmogenic cardiotoxicity of the quinoline and structurally related antimalarial drugs: A systematic review. BMC Med. 2018;16:200. PMC6220451.

Marmor MF, Kellner U, Lai TY, Lyons JS, Mieler WF; American Academy of Ophthalmology. Revised recommendations on screening for chloroquine and hydroxychloroquine retinopathy. Ophthalmology. 2011;118(2):415–422. doi:10.1016/j.ophtha.2010.11.017

Yao X, Ye F, Zhang M, et al. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) [published online ahead of print, 2020 Mar 9]. *Clin Infect Dis*. 2020;ciaa237. doi:10.1093/cid/ciaa237

Vitamin D reference: https://ods.od.nih.gov/factsheets/VitaminD-HealthProfessional/